CLINICAL TRIAL: NCT07378657
Title: Systematic Management Approach for Children and Adolescents With Orbital Lymphatic Malformation
Brief Title: Systematic Approach for Children With Orbital Malformation With Sirolimus Use
Acronym: sirolimus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, nihal hussien aly, associate professor of pediatrics -pediatric hematology and oncology unit, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU R 271/2025
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Orbital Lymphatic Malformation
Keywords: sirolimus; orbital lymphatic malformation
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: All Patients with symptomatic LM except complex type (Active Comparator): Group 1: All Patients with symptomatic lymphatic malformation except those with complex lymphatic malformation.They will be assigned to sclerotherpay .Local intralesional trancutaneous injection dose will be 0.6 mg / kg of bleomycin dissolved in the total volume of the lesion calculated from dimensions of orbital lesion in MRI orbit with contrast. Intralesional injection frequency will be guided by clinical response of the patients and imaging studies.If there is response clinically, injection will be continued every one month until there is no further response or if the lesion is reaching 75% of lesion size Or if there is no response from first injection.For lid and conjunctival components local injection will be for small , moderate and large lesions 2 IU, 4 IU, 6 IU respectively and further injection every month guided by lesion response.Less than 25% reduction will not receive further injection, if there is 25%- 50 % reduction injection will continue till reaching 75%
  Interventions: Procedure: Injection Sclerotherapy
- Group 2: Patients with complex LM or patients from group 1 if no response (Active Comparator): Patients assigned to sirolimus arm will be patients with A) Patients with symptomatic complex lymphatic malformation. B) Patients in group 1 if there is progression in lesion size or ineffective local therapy.
  Dose will be 0.8 mg/m2 twice daily orally for 6 months ,published literature for sirolimus' use in the pediatric population recommends a starting dose of sirolimus 1.6 mg/m2/day divided twice daily (10) with target trough level of 8-15 ng/ml will be done after 2 weeks from starting therapy
  Interventions: Drug: Sirolimus (Rapamune®)
- Group 3: A) Patients in group 1 or complex if there is concern for complications like hemorrhage, am (Active Comparator): Dose will be 0.8 mg/m2 twice daily orally for 6 months ,published literature for sirolimus' use in the pediatric population recommends a starting dose of sirolimus 1.6 mg/m2/day divided twice daily (10) with target trough level of 8-15 ng/ml will be done after 2 weeks from starting therapy
  Interventions: Other: both injection sclerotherapy and sirolimus

INTERVENTIONS:
Procedure: Injection Sclerotherapy — For group 1: They will be assigned to sclerotherpay .Local intralesional trancutaneous injection dose will be 0.6 mg / kg of bleomycin dissolved in the total volume of the lesion calculated from dimensions of orbital lesion in MRI orbit with contrast. Intralesional injection frequency will be guided by clinical response of the patients and imaging studies.If there is response clinically, injection will be continued every one month until there is no further response or if the lesion is reaching 75% of lesion size Or if there is no response from first injection.For lid and conjunctival components local injection will be for small , moderate and large lesions 2 IU, 4 IU, 6 IU respectively and further injection every month guided by lesion response.Less than 25% reduction will not receive further injection, if there is 25%- 50 % reduction injection will continue till reaching 75% or more clinical reduction in size
  Arms: Group 1: All Patients with symptomatic LM except complex type
Drug: Sirolimus (Rapamune®) — Dose will be 0.8 mg/m2 twice daily orally for 6 months ,published literature for sirolimus' use in the pediatric population recommends a starting dose of sirolimus 1.6 mg/m2/day divided twice daily (10) with target trough level of 8-15 ng/ml will be done after 2 weeks from starting therapy
  Arms: Group 2: Patients with complex LM or patients from group 1 if no response
Other: both injection sclerotherapy and sirolimus — They will be assigned to sclerotherpay .Local intralesional trancutaneous injection dose will be 0.6 mg / kg of bleomycin dissolved in the total volume of the lesion calculated from dimensions of orbital lesion in MRI orbit with contrast. Intralesional injection frequency will be guided by clinical response of the patients and imaging studies.If there is response clinically, injection will be continued every one month until there is no further response or if the lesion is reaching 75% of lesion size Or if there is no response from first injection.For lid and conjunctival components local injection will be for small , moderate and large lesions 2 IU, 4 IU, 6 IU respectively and further injection every month guided by lesion response.Less than 25% reduction will not receive further injection, if there is 25%- 50 % reduction injection will continue till reaching 75% or more clinical reduction in size sirolimus will be given in a dose of 0.8 mg per m2 twice daily .
  Arms: Group 3: A) Patients in group 1 or complex if there is concern for complications like hemorrhage, am

SUMMARY:
The goal of this interventional study is to Set a systematic management approach for orbital lymphatic malformation and to study the safety and efficacy of sirolimus in children and adolescents with orbital lymphatic malformation]. The main questions it aims to answer are:

[what is the safety of using sirolimus in patients with orbital lymphatic malformation]? [what is the efficacy of sirolimus in patients with orbital lymphatic malformation]? Participants will be divided into three groups based on their symptoms, extent and type of orbital lymphatic malformation Group 1 ( will receive injection sclerotherapy): All Patients with symptomatic lymphatic malformation except those with complex malformation , Group 2 (will receive sirolimus on 0.8 mg per m2 twice daily for 6 months ):A) Patients with symptomatic complex lymphatic malformation.

B) Patients in group 1 if there is progression in lesion size or ineffective local therapy Group 3 ( will receive both injection sclerotherapy and sirolimus):A) Patients in group 1 and patients with complex lymphatic malformation if there is concern for complications like hemorrhage, amblyopia and vision loss since diagnosis.

DETAILED DESCRIPTION:
This is an interventional study aiming at setting systematic approach for children and adolescents with orbital lymphatic malformation and to assess the safety and efficacy of sirolimus in patients with orbital lymphatic malformation Patients with lymphatic malformation will be subdivided according 4 grades, grade1 the size of the cyst, grade 2 the extension , grade 3 the angiogensis , grade 4 according to symptoms Grade 1:According to the size of cyst, Lymphatic malformation are divided into macrocystic (>2cm), microcystic(<2cm) and mixed cyst.Grade 2: According to the extension , lymphatic malformation are divided into superficial (presenting as a subcutaneous cyst); deep (having orbital infiltration);combined (superficial and deep components); complex (intracranial or head and neck infiltration) (10).

Grade 3: According to angiogensis, lymphatic malformation are divided into simple lympahtic malformation or combined with venous element or capillary malformation Grade 4 : According to symptoms , lymphatic malformation are divided into asympyomatic and symptomatic Patients will be assigned to available treatment modality either local control via injection sclerotherapy or surgery verus sirolimus orally either alone or combined with local control.

Group 1: All Patients with symptomatic lymphatic malformation except those with complex lymphatic malformation.They will be assigned to sclerotherpay .Local intralesional trancutaneous injection dose will be 0.6 mg / kg of bleomycin dissolved in the total volume of the lesion calculated from dimensions of orbital lesion in MRI orbit with contrast. Intralesional injection frequency will be guided by clinical response of the patients and imaging studies.If there is response clinically, injection will be continued every one month until there is no further response or if the lesion is reaching 75% of lesion size Or if there is no response from first injection.For lid and conjunctival components local injection will be for small , moderate and large lesions 2 IU, 4 IU, 6 IU respectively and further injection every month guided by lesion response.Less than 25% reduction will not receive further injection, if there is 25%- 50 % reduction injection will continue till reaching 75% or more clinical reduction in size (9) Group 2: Patients assigned to sirolimus arm will be patients with A) Patients with symptomatic complex lymphatic malformation. B) Patients in group 1 if there is progression in lesion size or ineffective local therapy.

Group 3 :Patients assigned to both modality from the start :

A) Patients in group 1 or complex if there is concern for complications like hemorrhage, amblyopia and vision loss since diagnosis.

Dose will be 0.8 mg/m2 twice daily orally for 6 months ,published literature for sirolimus' use in the pediatric population recommends a starting dose of sirolimus 1.6 mg/m2/day divided twice daily (10) with target trough level of 8-15 ng/ml will be done after 2 weeks from starting therapy , available containing tablets are rapimmune tablets (1 mg), tablets should not be crushed nor chew, or spilted, it should be taken in the same way either with food or without.Grapefruit juice reduces CYP3A4-mediated drug metabolism. Grapefruit juice must not be taken with or used for dilution of Rapamune .Immunosuppressants may affect response to vaccination.During treatment with sirolimus, vaccination may be less effective. The use of live vaccines should be avoided; live vaccines may include, but are not limited to, the following: measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid

All patients will be subjected to the detailed history with data at diagnosis collected from the filing system

1. Detailed medical history with special emphasis on:Demographic data , the presenting symptoms, the course of the disease, any complications like proptosis , pain , bleeding or cosmetic disfigurement.Treatment that will be received including sclerotherapy ( type of sclerosant agent, frequency, dose and response assessment), drug therapy (sirolimus including dose , drug level, side effects and response assessment)
2. Thorough clinical examination laying stress on:

   Physical examination for the site , the size , the colour, the consistency , the tenderness, systemic examination for associated anomalies was done. Blood pressure measurement for patients on siroloimus at each visit.
3. Laboratory investigations:

Complete blood count (CBC) before intervention and after 2 weeks from starting sirolimus then every 3 months while the patient is receiving it. Sirolomus level for patients who are assigned to sirolimus after 2 weeks from starting therapy and in case of progression or development of reported side effect.

Alanine transaminase , serum creatinine, lipid profile including (cholesterol and triglycerides) after 3 months and after 6 months from start of treatment in patient group on sirolimus.

1- Radiological assessment:

1- MRI orbit and brain vascular anomaly protocol (conventional pre contrast MRI and dynamic post contrast sequences) to confirm diagnosis, and detect extension for deeper lesion and after 6 months of intervention to assess radiological improvement.

ELIGIBILITY:
Inclusion Criteria:

Age : 1-18 years Children and adolescents diagnosed with orbital low flow vascular malformation based on clinical , radilogical findings

Exclusion Criteria:

Children and adolescents with orbital high flow vascular malformation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
safety of sirolimus in patients with orbital lymphatic malformation | 6 months
  assessment of safety of sirolimus

SECONDARY OUTCOMES:
efficacy of sirolimus in patients with orbital malformation | 6 months
  reduction size of the lymphatic malformation and recovery of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available upon request